CLINICAL TRIAL: NCT00379561
Title: A Phase 1 Trial of PSA-Activated PSA-PAH1 Therapy for Locally Recurrent Prostate Cancer Without Metastases After Primary Radiation Therapy
Brief Title: PSA-Activated PSA-PAH1 for Locally Recurrent Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sophiris Bio Corp (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PRX302
Record Dates: First submitted 2006-09-20; First posted 2006-09-22 (Estimated); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Recurrent Prostate Cancer; Non-Metastatic prostate cancer; Recurrent Localized Prostate Cancer with Biochemical Failure
MeSH Terms: conditions — Prostatic Neoplasms | interventions — PRX302

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Intervention PSA-PAH1 (Experimental): Determination of the therapeutic activity of different concentrations of PSA-PAH1 at increasing doses of per gram of prostate.
  Interventions: Drug: PSA-Activated PSA-PAH1

INTERVENTIONS:
Drug: PSA-Activated PSA-PAH1
  Other Names: PRX302, Topsalysin

SUMMARY:
This Phase 1 trial will evaluate the safety and tolerability of PSA-Activated PSA-PAH1 in subjects who have shown biochemical failure and have either completed at least one primary radiation therapy for prostate cancer and have evidence of recurrent local prostate cancer without metastases.

DETAILED DESCRIPTION:
For more information please contact Primary Investigator or Protox Therapeutics, Inc.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Histologically proven prostate adenocarcinoma
* Completed a full course of definitive external beam radiation or definitive brachytherapy (but not both) as primary therapy for diagnosed prostate cancer at least one year prior to enrollment
* Subject must have at least one available PSA measurement that was taken 60 days or more following their primary therapy, but no later than 2 months prior to their screening visit (this measurement will serve as the first time point for computing a screening value for PSA doubling time)
* Subject's PSA doubling time at screening must be > 3 months (this doubling time will be computed by comparing the earliest available PSA that is 60 days or more following the subject's primary therapy but no later than 2 months prior to their screening visit, to the PSA measurement obtained during the screening visit)
* Within one year prior to enrollment:

  * Demonstrated "biochemical failure," as determined by three consecutive increases in PSA at least 2 weeks apart
  * Multiple-site biopsy-confirmed local recurrence of prostate cancer
* Within 3 months prior to enrollment:

  * No evidence of metastatic disease including no bone metastases on bone scan, or any lymph node, lung, liver or soft tissue metastases on a CT or MRI scan or any other evidence of metastatic disease
  * No receipt of androgen ablation therapy [Note: Subjects may have received androgen ablation therapy in the past, but not within 3 months prior to enrollment. No subject will be removed from androgen ablation therapy prior to this trial to permit/facilitate eligibility for this trial.]
* Within 30 days prior to enrollment:

  * Prostate gland weighing less than 40 g estimated on the basis of CT/ultrasound data
  * Serum testosterone above castrate range (> 1 ng/dL)
  * PSA level less than 20 ng/mL
  * Eastern Cooperative Oncology Group (ECOG) score of 0-2
  * Written informed consent
  * Adequate organ function as evidenced by:

Exclusion Criteria:

* Any history of active malignancy other than prostate cancer
* Have active viral, bacterial or fungal infections that require systemic therapy
* Prior biological, immunological or chemotherapy for prostate cancer
* Receiving concurrent medication for prostate cancer
* Received as primary therapy for prostate cancer, definitive external beam radiation and concomitant brachytherapy
* Prior history of metastatic prostate cancer
* Treatment with other investigational therapies within 12 months prior to enrollment that could produce a compromised immune system, or receipt of immunosuppressive drugs including corticosteroids or ketoconazole within 1 month prior to enrollment, or a history of immunodeficiency disease
* Recurrence of prostate cancer within 6 months after initiation of primary radiotherapy
* Active heart, liver, lung, renal disease, active infection or other serious uncontrolled illnesses
* Positive antibody test during screening for HIV-1, HIV-2, HTLV-1, HTLV-2, Hep B, or Hep C
* Unable or unwilling to return for required visits and follow-up examinations
* Have a chronic indwelling Foley catheter for obstructive uropathy
* Received salvage external beam radiotherapy and/or salvage seed brachytherapy prior to enrollment
* Received prior treatment with PSA-PAH1 (subjects may not be redosed under this protocol)
* Men unwilling to use condoms for the duration of the study (3 months) to prevent a pregnancy, and to avoid semen contact with their partner.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2006-03; Primary Completion 2007-05 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerance of PSA-PAH1
MTD of PSA-PAH1

SECONDARY OUTCOMES:
Pharmacokinetic data on PSA-PAH1
Immune response to PSA-PAH1
Evidence of activity of PSA-PAH1

CONTACTS AND LOCATIONS:
Overall Officials: King S Coffield, M.D., Principal Investigator — Cancer Research Institute of Scott and White
Locations (1):
- Cancer Research Institute of Scott and White, Temple, Texas, United States